CLINICAL TRIAL: NCT05293236
Title: A Double Blind, Placebo-Controlled, Randomized, Phase Ib Clinical Study of ApTOLL for the Treatment of COVID-19
Brief Title: ApTOLL for the Treatment of COVID-19
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Lack of patients due to reduced incidence in the COVID-19 infected population in Spain
Sponsor: Macarena Hernández Jiménez (Industry)
Collaborators: Centro para el Desarrollo Tecnológico Industrial (Unknown)
Responsible Party: Sponsor-Investigator, Macarena Hernández Jiménez, PhD, aptaTargets S.L.
Organization: aptaTargets S.L. (Industry)
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: APTACOVID
Record Dates: First submitted 2022-03-18; First posted 2022-03-24 (Actual); Last update posted 2023-08-07 (Actual); Status verified 2023-08

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — TLR4 antagonist ApTOLL; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Placebo (Placebo Comparator): Nine COVID-19 patients (three from each treatment-group) treated with saline intravenous infusion
  Interventions: Other: Saline
- Dose 1 (Experimental): Seven COVID-19 patients treated with ApTOLL (0.05mg/kg) intravenous infusion
  Interventions: Drug: ApTOLL
- Dose 2 (Experimental): Seven COVID-19 patients treated with ApTOLL (0.1mg/kg) intravenous infusion
  Interventions: Drug: ApTOLL
- Dose 3 (Experimental): Seven COVID-19 patients treated with ApTOLL (0.2mg/kg) intravenous infusion
  Interventions: Drug: ApTOLL

INTERVENTIONS:
Drug: ApTOLL — ApTOLL is an aptamer (DNA single strain) designed to block TLR4 (toll-like receptor 4)
  Arms: Dose 1; Dose 2; Dose 3
Other: Saline — Saline for intravenous infusion
  Arms: Placebo

SUMMARY:
There is a clear and urgent medical need of developing new medicinal products for COVID-19 since there are poor pharmacological tools to block the progression of patients to cytokine storm syndrome (CSS). To this aim, this Phase Ib clinical study (APTACOVID) pretends to determine whether ApTOLL, in combination with the standard of care, is safe and shows any biological effect) in those patients infected with SARS-CoV-2 who are not developed CSS yet.

ELIGIBILITY:
Inclusion Criteria:

1. Men or women with age ≥18 and ≤85 years.
2. In case of women of childbearing potential (WOCBP), they should confirm menstrual period and a negative highly sensitive urine or serum pregnancy test to be included.
3. Laboratory-confirmed SARS-CoV-2 infection.
4. Informed consent obtained .
5. Hypoxia (SpO2<95%).
6. Documented lung opacities/infiltrates.
7. Confirmed hyperinflammation.

Exclusion Criteria:

1. Onset of symptoms of COVID-19 >14 days.
2. Pregnant or nursing (lactating) women.
3. Hospitalized >10 days for COVID-19.
4. Need of high concentration non-rebreather mask, high-flow nasal cannula , non-invasive mechanical ventilation or invasive mechanical ventilation.
5. Systolic blood pressure < 90 mmHg.
6. Serious concomitant illness.
7. Recent treatment with cell-depleting therapies.
8. Enrolled in another clinical trial.
9. Severe renal dysfunction.
10. In the opinion of the investigator, unable to comply with the requirements to participate in the study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2022-01-14 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Incidence of Death | From dosing to day 28 after administration
  Number of dead patients at the end of the study
Incidence of Adverse Events as assessed by MedDRA | From dosing to day 28 after administration
  Adverse events that occur during the study
Number of patients with treatment-related alterations coagulation parameters | From dosing to day 28 after administration
  Protrombine Time (PT) and activated Partial Tromboplastine Time (aPTT)
Number of patients with treatment-related alterations Complement Factors | From dosing to day 28 after administration
  Complement activation determined in blood

CONTACTS AND LOCATIONS:
Overall Officials: Macarena Hernández, PhD, Study Director — aptaTargets S.L.; Sergio Serrano, MD, Principal Investigator — Hospital Universitario Ramón y Cajal; Ignacio Santos, MD, Principal Investigator — Hospital Universitario La Princesa; Marc Ribó, MD, PhD, Study Director — aptaTargets S.L.
Locations (4):
- Spain (4):
  - Hospital Universitario de Burgos, Burgos
  - Hospital Universitario Clínico San Carlos, Madrid
  - Hospital Universitario La Princesa, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid

IPD SHARING:
Plan to Share IPD: Undecided
We have not planned this point yet

REFERENCES:
- See also: Related Info — http://aptatargets.com